CLINICAL TRIAL: NCT03040388
Title: Predicting Effects and Risk of Relapse Into Depression - The Danish ECT/MRI Project
Brief Title: Exploring Effects of Electroconvulsive Therapy on the Human Brain in Depression - The Danish ECT/MRI Study
Status: Completed | Type: Observational
Sponsor: University of Copenhagen (Other)
Collaborators: Glostrup University Hospital, Copenhagen (Other); Amager Hospital (Other); Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Responsible Party: Principal Investigator, Poul Videbech, Professor, consultant in psychiatry, University of Copenhagen
Other Study IDs: DK-ECT-MR-1
Record Dates: First submitted 2017-01-30; First posted 2017-02-02 (Estimated); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Depressive Disorder; Depression; Depressive Disorder, Major
Keywords: Electroconvulsive therapy; Depressive Disorder; Magnetic Resonance Imaging; Hippocampus; Brain-Derived Neurotrophic Factor; Vascular Endothelial Growth Factor; Blood-Brain Barrier
MeSH Terms: conditions — Depressive Disorder; Depression; Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples are kept in the biobank until the last enrolled patient has been examined. They will be then analysed for S100B-protein concentration and destroyed. Whole blood, serum and plasma samples are kept in the biobank until the last enrolled patient has been examined. They will then be analysed for concentrations of BDNF and VEGF and destroyed. Extra whole blood samples are stored in the psychiatric biobank for the future research (as part of another protocol - PSV-2001-04, I-Suite 00422 - ID nr 2001-54-798)
Oversight: Data Monitoring Committee: No

SUMMARY:
The main purpose of this study is to determine whether electroconvulsive therapy (ECT) causes any structural or functional brain changes and thus indicating its mechanism of action. The second aim is to find predictors of an immediate response, sustained remission, relapse and side-effects. Thirdly, this study aims to explore whether ECT causes any changes in blood-brain barriers permeability and whether these changes correlate to memory problems. The fourth objective is to examine whether ECT causes any brain tissue damage.

DETAILED DESCRIPTION:
ECT has been the most effective treatment of depression for decades. Despite of this, neither the mechanism of action or side-effects are fully elucidated. The reason why some patients relapse shortly after remission is still not completely understood. Thus, there is a need to find predictors of the favourable clinical effect, relapse and side-effects. ECT is considered by professionals to be a safe procedure. However, this view is based on rather old and small studies. Additionally, many patients do not consent to this treatment because they fear a permanent loss of memory or that they will contract a brain damage after the completed ECT series. Therefore, it is very important to examine whether ECT might have negative effects on the structure or function of the brain, using state of the art Magnetic Resonance Imaging (MRI) techniques on a greater study population.

The study consists of 60 inpatients, diagnosed with depression, admitted to one of the recruiting Mental Health Centres, and scheduled to ECT. The most modern MRI sequences examining brain structure and function are used at 3 time points: at baseline (just before ECT series), the second examination (just after ECT series) and the third (follow-up) examination (6 months after ECT series). Blood samples (measurements of Brain-Derived Neurotrophic Factor - BDNF, Vascular Endothelial Growth Factor - VEGF along with the marker of brain injury - S100B-protein) and the evaluation of clinical effect and side-effects to ECT are performed at the same time points.

The study has 4 main hypotheses. The first hypothesis assumes that the immediate and sustained response to ECT can be predicted by combining neuroimaging findings and blood-samples results. The second hypothesis is based on the assumption that ECT modulates the microstructure and connectivity in the fronto-limbic pathways (FLPs) and that this modulation correlates with the clinical effect. Thus, the altered microstructure of the FLPs in depression is normalised by an ECT series. Furthermore, the depression-associated increased resting state connectivity in FLPs is normalised by ECT. The third hypothesis is that ECT will induce changes in blood-brain barrier (BBB) permeability, which will correlate with the severity of memory problems. The last hypothesis assumes that ECT does not cause any brain tissue damage (including brain atrophy and white matter lesions - WMLs).

ELIGIBILITY:
Inclusion Criteria:

* age 18-95 years
* admitted at the MHC Glostrup, MHC Amager or MHC Copenhagen (or other Mental Health Centres in the Capital Region)
* fulfilling the criteria for depression according to ICD-10 and major depression according to DSM-IV and where ECT is planned.
* must be able to give informed consent to participate in the study

Exclusion Criteria:

* Schizophrenia or any other psychotic disorder except for psychotic depression
* Dependency syndrome according to ICD-10.
* Severe somatic or neurological condition (e.g. stroke) confounding results
* Head trauma resulting in unconsciousness for more than 5 minutes
* Severe psychotic symptoms or suicide impulses making transportation hazardous
* Contraindications against MRI or Gadovist infusion
* Pregnancy
* Maintenance ECT or ECT received during the last 6 months
* Any form of compulsory treatment
* Subjects who do not consent to be informed of incidental findings that could have healthcare implications will not be scanned and can thus not be included

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of the inpatients admitted to one of the recruiting Mental Health Centres (MHC) in the Capital Region of Denmark (Mental Health Centre Glostrup or Amager or Copenhagen or others), diagnosed with either depression according to the 10th version of the International Classification of Diseases (ICD-10) or major depression according to the Diagnostic and Statistical Manual of Mental Disorders, 4th ed (DSM-IV) and scheduled to ECT series.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2017-08-09 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2020-06-11 (Actual)

PRIMARY OUTCOMES:
Volumetric changes in the hippocampus. | at 3 time points: at baseline (before ECT series), after an ECT series (+3 day), at follow-up (6 months after the ECT series)
  This outcome will be measured by means of voxel-based morphometry (VBM).
Changes in BDNF concentration in the blood. | at 3 time points: at baseline (before ECT series), after an ECT series (+3 day), at follow-up (6 months after the ECT series)
Changes in regional cerebral blood flow (rCBF) in the frontal lobes. | at 3 time points: at baseline (before ECT series), after an ECT series (+3 day), at follow-up (6 months after the ECT series)
  Pseudo-continuous arterial spin-labelling (PSCAL) will be used to measure this outcome.

SECONDARY OUTCOMES:
The number of WMLs in the brain. | at 3 time points: at baseline (before ECT series), after an ECT series (+3 day), at follow-up (6 months after the ECT series)
  FLAIR sequences of MRI will be used to measure this outcome.
Changes in water diffusion in the brain. | at 3 time points: at baseline (before ECT series), after an ECT series (+3 day), at follow-up (6 months after the ECT series)
  Diffusion-weighted imaging (DWI) will be used to measure this outcome.
Changes in the level of fractional anisotropy (FA) in the brain. | at 3 time points: at baseline (before ECT series), after an ECT series (+3 day), at follow-up (6 months after the ECT series)
  Diffusion tensor imaging (DTI) will be used to measure this outcome.
Changes in the level of intrinsic connectivity pattern in fronto-limbic pathways in the brain. | at 3 time points: at baseline (before ECT series), after an ECT series (+3 day), at follow-up (6 months after the ECT series)
  Resting state functional MRI will be used to measure this outcome.
Changes in the glucose metabolism in the brain. | at 3 time points: at baseline (before ECT series), after an ECT series (+3 day), at follow-up (6 months after the ECT series)
  Cerebral Metabolic Rate of Oxygen ( CMRO2) will be used to measure this outcome.
Changes in blood-brain barrier (BBB) permeability. | at 3 time points: at baseline (before ECT series), after an ECT series (+3 day), at follow-up (6 months after the ECT series)
  Dynamic Contrast Enhanced (DCE)T1-weighted imaging will be used to measure this outcome.
Changes in S100B-protein concentration in the blood. | at 3 time points: at baseline (before ECT series), after an ECT series (+3 day), at follow-up (6 months after the ECT series)

CONTACTS AND LOCATIONS:
Overall Officials: Poul Videbech, Professor, Principal Investigator — Glostrup University Hospital, Copenhagen
Locations (1):
- Mental Health Centre Glostrup, Glostrup Municipality, The Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No
There is no plan to share Individual Patient Data.

REFERENCES:
- [Background] Abbott CC, Gallegos P, Rediske N, Lemke NT, Quinn DK. A review of longitudinal electroconvulsive therapy: neuroimaging investigations. J Geriatr Psychiatry Neurol. 2014 Mar;27(1):33-46. doi: 10.1177/0891988713516542. Epub 2013 Dec 30. PMID 24381234
- [Background] Andrade C, Bolwig TG. Electroconvulsive therapy, hypertensive surge, blood-brain barrier breach, and amnesia: exploring the evidence for a connection. J ECT. 2014 Jun;30(2):160-4. doi: 10.1097/YCT.0000000000000133. PMID 24800688
- [Background] Ahdidan J, Hviid LB, Chakravarty MM, Ravnkilde B, Rosenberg R, Rodell A, Stodkilde-Jorgensen H, Videbech P. Longitudinal MR study of brain structure and hippocampus volume in major depressive disorder. Acta Psychiatr Scand. 2011 Mar;123(3):211-9. doi: 10.1111/j.1600-0447.2010.01644.x. Epub 2011 Jan 11. PMID 21219263
- [Background] Arts B, Peters M, Ponds R, Honig A, Menheere P, van Os J. S100 and impact of ECT on depression and cognition. J ECT. 2006 Sep;22(3):206-12. doi: 10.1097/01.yct.0000235925.37494.2c. PMID 16957538
- [Background] Awata S, Konno M, Kawashima R, Suzuki K, Sato T, Matsuoka H, Fukuda H, Sato M. Changes in regional cerebral blood flow abnormalities in late-life depression following response to electroconvulsive therapy. Psychiatry Clin Neurosci. 2002 Feb;56(1):31-40. doi: 10.1046/j.1440-1819.2002.00927.x. PMID 11929569
- [Background] Bergsholm P, Larsen JL, Rosendahl K, Holsten F. Electroconvulsive therapy and cerebral computed tomography. A prospective study. Acta Psychiatr Scand. 1989 Dec;80(6):566-72. doi: 10.1111/j.1600-0447.1989.tb03027.x. PMID 2618780
- [Background] Beyer JL. Volumetric brain imaging studies in the elderly with mood disorders. Curr Psychiatry Rep. 2006 Feb;8(1):18-24. doi: 10.1007/s11920-006-0077-0. PMID 16513039
- [Background] Bolwig TG, Hertz MM, Paulson OB, Spotoft H, Rafaelsen OJ. The permeability of the blood-brain barrier during electrically induced seizures in man. Eur J Clin Invest. 1977 Apr;7(2):87-93. doi: 10.1111/j.1365-2362.1977.tb01578.x. PMID 404164
- [Background] Bolwig TG. How does electroconvulsive therapy work? Theories on its mechanism. Can J Psychiatry. 2011 Jan;56(1):13-8. doi: 10.1177/070674371105600104. PMID 21324238
- [Background] Bolwig TG. Neuroimaging and electroconvulsive therapy: a review. J ECT. 2014 Jun;30(2):138-42. doi: 10.1097/YCT.0000000000000140. PMID 24800687
- [Background] Bronge L, Wahlund LO. White matter changes in dementia: does radiology matter? Br J Radiol. 2007 Dec;80 Spec No 2:S115-20. doi: 10.1259/bjr/35265137. PMID 18445741
- [Background] Brunoni AR, Baeken C, Machado-Vieira R, Gattaz WF, Vanderhasselt MA. BDNF blood levels after electroconvulsive therapy in patients with mood disorders: a systematic review and meta-analysis. World J Biol Psychiatry. 2014 Jul;15(5):411-8. doi: 10.3109/15622975.2014.892633. Epub 2014 Mar 16. PMID 24628093
- [Background] Campbell JJ 3rd, Coffey CE. Neuropsychiatric significance of subcortical hyperintensity. J Neuropsychiatry Clin Neurosci. 2001 Spring;13(2):261-88. doi: 10.1176/jnp.13.2.261. No abstract available. PMID 11449035
- [Background] Coffey CE, Weiner RD, Djang WT, Figiel GS, Soady SA, Patterson LJ, Holt PD, Spritzer CE, Wilkinson WE. Brain anatomic effects of electroconvulsive therapy. A prospective magnetic resonance imaging study. Arch Gen Psychiatry. 1991 Nov;48(11):1013-21. doi: 10.1001/archpsyc.1991.01810350053008. PMID 1747016
- [Background] Dukart J, Regen F, Kherif F, Colla M, Bajbouj M, Heuser I, Frackowiak RS, Draganski B. Electroconvulsive therapy-induced brain plasticity determines therapeutic outcome in mood disorders. Proc Natl Acad Sci U S A. 2014 Jan 21;111(3):1156-61. doi: 10.1073/pnas.1321399111. Epub 2013 Dec 30. PMID 24379394
- [Background] Fitzgerald PB, Laird AR, Maller J, Daskalakis ZJ. A meta-analytic study of changes in brain activation in depression. Hum Brain Mapp. 2008 Jun;29(6):683-95. doi: 10.1002/hbm.20426. PMID 17598168
- [Background] UK ECT Review Group. Efficacy and safety of electroconvulsive therapy in depressive disorders: a systematic review and meta-analysis. Lancet. 2003 Mar 8;361(9360):799-808. doi: 10.1016/S0140-6736(03)12705-5. PMID 12642045
- [Background] Herrmann LL, Le Masurier M, Ebmeier KP. White matter hyperintensities in late life depression: a systematic review. J Neurol Neurosurg Psychiatry. 2008 Jun;79(6):619-24. doi: 10.1136/jnnp.2007.124651. Epub 2007 Aug 23. PMID 17717021
- [Background] Jorgensen A, Magnusson P, Hanson LG, Kirkegaard T, Benveniste H, Lee H, Svarer C, Mikkelsen JD, Fink-Jensen A, Knudsen GM, Paulson OB, Bolwig TG, Jorgensen MB. Regional brain volumes, diffusivity, and metabolite changes after electroconvulsive therapy for severe depression. Acta Psychiatr Scand. 2016 Feb;133(2):154-164. doi: 10.1111/acps.12462. Epub 2015 Jul 3. PMID 26138003
- [Background] Joshi SH, Espinoza RT, Pirnia T, Shi J, Wang Y, Ayers B, Leaver A, Woods RP, Narr KL. Structural Plasticity of the Hippocampus and Amygdala Induced by Electroconvulsive Therapy in Major Depression. Biol Psychiatry. 2016 Feb 15;79(4):282-92. doi: 10.1016/j.biopsych.2015.02.029. Epub 2015 Mar 5. PMID 25842202
- [Background] Kho KH, van Vreeswijk MF, Simpson S, Zwinderman AH. A meta-analysis of electroconvulsive therapy efficacy in depression. J ECT. 2003 Sep;19(3):139-47. doi: 10.1097/00124509-200309000-00005. PMID 12972983
- [Background] Kranaster L, Janke C, Mindt S, Neumaier M, Sartorius A. Protein S-100 and neuron-specific enolase serum levels remain unaffected by electroconvulsive therapy in patients with depression. J Neural Transm (Vienna). 2014 Nov;121(11):1411-5. doi: 10.1007/s00702-014-1228-9. Epub 2014 May 7. PMID 24801966
- [Background] Li CT, Lin CP, Chou KH, Chen IY, Hsieh JC, Wu CL, Lin WC, Su TP. Structural and cognitive deficits in remitting and non-remitting recurrent depression: a voxel-based morphometric study. Neuroimage. 2010 Mar;50(1):347-56. doi: 10.1016/j.neuroimage.2009.11.021. Epub 2009 Nov 26. PMID 19931620
- [Background] Lyden H, Espinoza RT, Pirnia T, Clark K, Joshi SH, Leaver AM, Woods RP, Narr KL. Electroconvulsive therapy mediates neuroplasticity of white matter microstructure in major depression. Transl Psychiatry. 2014 Apr 8;4(4):e380. doi: 10.1038/tp.2014.21. PMID 24713861
- [Background] Mander AJ, Whitfield A, Kean DM, Smith MA, Douglas RH, Kendell RE. Cerebral and brain stem changes after ECT revealed by nuclear magnetic resonance imaging. Br J Psychiatry. 1987 Jul;151:69-71. doi: 10.1192/bjp.151.1.69. PMID 3676627
- [Background] Menken M, Safer J, Goldfarb C, Varga E. Multiple ECT: morphologic effects. Am J Psychiatry. 1979 Apr;136(4A):453. No abstract available. PMID 426115
- [Background] Najjar S, Pearlman DM, Devinsky O, Najjar A, Zagzag D. Neurovascular unit dysfunction with blood-brain barrier hyperpermeability contributes to major depressive disorder: a review of clinical and experimental evidence. J Neuroinflammation. 2013 Dec 1;10:142. doi: 10.1186/1742-2094-10-142. PMID 24289502
- [Background] Nobler MS, Oquendo MA, Kegeles LS, Malone KM, Campbell CC, Sackeim HA, Mann JJ. Decreased regional brain metabolism after ect. Am J Psychiatry. 2001 Feb;158(2):305-8. doi: 10.1176/appi.ajp.158.2.305. PMID 11156816
- [Background] Nobuhara K, Okugawa G, Minami T, Takase K, Yoshida T, Yagyu T, Tajika A, Sugimoto T, Tamagaki C, Ikeda K, Sawada S, Kinoshita T. Effects of electroconvulsive therapy on frontal white matter in late-life depression: a diffusion tensor imaging study. Neuropsychobiology. 2004;50(1):48-53. doi: 10.1159/000077941. PMID 15179020
- [Background] Nordanskog P, Dahlstrand U, Larsson MR, Larsson EM, Knutsson L, Johanson A. Increase in hippocampal volume after electroconvulsive therapy in patients with depression: a volumetric magnetic resonance imaging study. J ECT. 2010 Mar;26(1):62-7. doi: 10.1097/YCT.0b013e3181a95da8. PMID 20190603
- [Background] Pagnin D, de Queiroz V, Pini S, Cassano GB. Efficacy of ECT in depression: a meta-analytic review. J ECT. 2004 Mar;20(1):13-20. doi: 10.1097/00124509-200403000-00004. PMID 15087991
- [Background] Palmio J, Huuhka M, Laine S, Huhtala H, Peltola J, Leinonen E, Suhonen J, Keranen T. Electroconvulsive therapy and biomarkers of neuronal injury and plasticity: Serum levels of neuron-specific enolase and S-100b protein. Psychiatry Res. 2010 May 15;177(1-2):97-100. doi: 10.1016/j.psychres.2009.01.027. Epub 2010 Apr 8. PMID 20378182
- [Background] Perrin JS, Merz S, Bennett DM, Currie J, Steele DJ, Reid IC, Schwarzbauer C. Electroconvulsive therapy reduces frontal cortical connectivity in severe depressive disorder. Proc Natl Acad Sci U S A. 2012 Apr 3;109(14):5464-8. doi: 10.1073/pnas.1117206109. Epub 2012 Mar 19. PMID 22431642
- [Background] Puri BK, Oatridge A, Saeed N, Ging JE, McKee HM, Lekh SK, Hajnal JV. Does electroconvulsive therapy lead to changes in cerebral structure. Br J Psychiatry. 1998 Sep;173:267. doi: 10.1192/bjp.173.3.267a. No abstract available. PMID 9926105
- [Background] Rocha RB, Dondossola ER, Grande AJ, Colonetti T, Ceretta LB, Passos IC, Quevedo J, da Rosa MI. Increased BDNF levels after electroconvulsive therapy in patients with major depressive disorder: A meta-analysis study. J Psychiatr Res. 2016 Dec;83:47-53. doi: 10.1016/j.jpsychires.2016.08.004. Epub 2016 Aug 5. PMID 27552533
- [Background] Sackeim HA. The anticonvulsant hypothesis of the mechanisms of action of ECT: current status. J ECT. 1999 Mar;15(1):5-26. PMID 10189616
- [Background] Scott AI, Douglas RH, Whitfield A, Kendell RE. Time course of cerebra; magnetic resonance changes after electroconvulsive therapy. Br J Psychiatry. 1990 Apr;156:551-3. doi: 10.1192/bjp.156.4.551. PMID 2386865
- [Background] Semkovska M, McLoughlin DM. Objective cognitive performance associated with electroconvulsive therapy for depression: a systematic review and meta-analysis. Biol Psychiatry. 2010 Sep 15;68(6):568-77. doi: 10.1016/j.biopsych.2010.06.009. Epub 2010 Jul 31. PMID 20673880
- [Background] Semkovska M, McLoughlin DM. Measuring retrograde autobiographical amnesia following electroconvulsive therapy: historical perspective and current issues. J ECT. 2013 Jun;29(2):127-33. doi: 10.1097/YCT.0b013e318279c2c9. PMID 23303426
- [Background] Shalev H, Serlin Y, Friedman A. Breaching the blood-brain barrier as a gate to psychiatric disorder. Cardiovasc Psychiatry Neurol. 2009;2009:278531. doi: 10.1155/2009/278531. Epub 2009 Aug 27. PMID 19936105
- [Background] Sheline YI, Price JL, Yan Z, Mintun MA. Resting-state functional MRI in depression unmasks increased connectivity between networks via the dorsal nexus. Proc Natl Acad Sci U S A. 2010 Jun 15;107(24):11020-5. doi: 10.1073/pnas.1000446107. Epub 2010 Jun 1. PMID 20534464
- [Background] Stelzhammer V, Rothermundt M, Guest PC, Michael N, Sondermann C, Kluge W, Martins-de-Souza D, Rahmoune H, Bahn S. Proteomic changes induced by anaesthesia and muscle relaxant treatment prior to electroconvulsive therapy. Proteomics Clin Appl. 2011 Dec;5(11-12):644-9. doi: 10.1002/prca.201100040. PMID 22006837
- [Background] Szabo K, Hirsch JG, Krause M, Ende G, Henn FA, Sartorius A, Gass A. Diffusion weighted MRI in the early phase after electroconvulsive therapy. Neurol Res. 2007 Apr;29(3):256-9. doi: 10.1179/174313206X153842. PMID 17509223
- [Background] Takano H, Motohashi N, Uema T, Ogawa K, Ohnishi T, Nishikawa M, Kashima H, Matsuda H. Changes in regional cerebral blood flow during acute electroconvulsive therapy in patients with depression: positron emission tomographic study. Br J Psychiatry. 2007 Jan;190:63-8. doi: 10.1192/bjp.bp.106.023036. PMID 17197658
- [Background] Taylor SM. Electroconvulsive therapy, brain-derived neurotrophic factor, and possible neurorestorative benefit of the clinical application of electroconvulsive therapy. J ECT. 2008 Jun;24(2):160-5. doi: 10.1097/YCT.0b013e3181571ad0. PMID 18580563
- [Background] Ten Doesschate F, van Eijndhoven P, Tendolkar I, van Wingen GA, van Waarde JA. Pre-treatment amygdala volume predicts electroconvulsive therapy response. Front Psychiatry. 2014 Nov 26;5:169. doi: 10.3389/fpsyt.2014.00169. eCollection 2014. PMID 25505429
- [Background] Tendolkar I, van Beek M, van Oostrom I, Mulder M, Janzing J, Voshaar RO, van Eijndhoven P. Electroconvulsive therapy increases hippocampal and amygdala volume in therapy refractory depression: a longitudinal pilot study. Psychiatry Res. 2013 Dec 30;214(3):197-203. doi: 10.1016/j.pscychresns.2013.09.004. Epub 2013 Oct 3. PMID 24090511
- [Background] Videbech P. MRI findings in patients with affective disorder: a meta-analysis. Acta Psychiatr Scand. 1997 Sep;96(3):157-68. doi: 10.1111/j.1600-0447.1997.tb10146.x. PMID 9296545
- [Background] Videbech P. PET measurements of brain glucose metabolism and blood flow in major depressive disorder: a critical review. Acta Psychiatr Scand. 2000 Jan;101(1):11-20. doi: 10.1034/j.1600-0447.2000.101001011.x. PMID 10674946
- [Background] Videbech P, Ravnkilde B, Pedersen AR, Egander A, Landbo B, Rasmussen NA, Andersen F, Stodkilde-Jorgensen H, Gjedde A, Rosenberg R. The Danish PET/depression project: PET findings in patients with major depression. Psychol Med. 2001 Oct;31(7):1147-58. doi: 10.1017/s0033291701004469. PMID 11681541
- [Background] Videbech P, Ravnkilde B, Pedersen TH, Hartvig H, Egander A, Clemmensen K, Rasmussen NA, Andersen F, Gjedde A, Rosenberg R. The Danish PET/depression project: clinical symptoms and cerebral blood flow. A regions-of-interest analysis. Acta Psychiatr Scand. 2002 Jul;106(1):35-44. doi: 10.1034/j.1600-0447.2002.02245.x. PMID 12100346
- [Background] Videbech P, Ravnkilde B. Hippocampal volume and depression: a meta-analysis of MRI studies. Am J Psychiatry. 2004 Nov;161(11):1957-66. doi: 10.1176/appi.ajp.161.11.1957. PMID 15514393
- [Background] Videbech P, Tehrani ES. [Imaging techniques and proposed implementation of a neuropsychiatric assessment program for patients with depression]. Ugeskr Laeger. 2007 Apr 16;169(16):1431-4. Danish. PMID 17484837
- [Background] Zachrisson OC, Balldin J, Ekman R, Naesh O, Rosengren L, Agren H, Blennow K. No evident neuronal damage after electroconvulsive therapy. Psychiatry Res. 2000 Oct 30;96(2):157-65. doi: 10.1016/s0165-1781(00)00202-x. PMID 11063788
- [Background] Zimmermann R, Schmitt H, Rotter A, Sperling W, Kornhuber J, Lewczuk P. Transient increase of plasma concentrations of amyloid beta peptides after electroconvulsive therapy. Brain Stimul. 2012 Jan;5(1):25-9. doi: 10.1016/j.brs.2011.01.007. Epub 2011 Mar 12. PMID 22037136
- [Derived] Gbyl K, Rostrup E, Raghava JM, Carlsen JF, Schmidt LS, Lindberg U, Ashraf A, Jorgensen MB, Larsson HBW, Rosenberg R, Videbech P. Cortical thickness following electroconvulsive therapy in patients with depression: a longitudinal MRI study. Acta Psychiatr Scand. 2019 Sep;140(3):205-216. doi: 10.1111/acps.13068. PMID 31265120
- [Derived] Saricicek Aydogan A, Oztekin E, Esen ME, Dusmez S, Gelal F, Besiroglu L, Zorlu N. Cortical thickening in remitters compared to non-remitters with major depressive disorder following 8-week antidepressant treatment. Acta Psychiatr Scand. 2019 Sep;140(3):217-226. doi: 10.1111/acps.13065. Epub 2019 Jul 17. PMID 31250445
- See also: Sundhedsstyrelsen: Referenceprogram for Unipolar Depression hos voksne. 2007. — http://www.sst.dk/~/media/6F9CE14B6FF245AABCD222575787FEB7.ashx
- See also: Ottosson J-O, Fink M. Ethics in electroconvulsive therapy. New York: Brunner-Reoutledge, 2004. — http://www.amazon.com/Ethics-Electroconvulsive-Therapy-Jan-Otto-Ottosson/dp/041594659X